CLINICAL TRIAL: NCT01450540
Title: Automated Graduated CPAP (AGPAP) for Improved Adherence in Newly Diagnosed OSA Patients: Multicenter Trial
Brief Title: Automated Graduated CPAP (AGPAP) for Improved Adherence in Newly Diagnosed Obstructive Sleep Apnea (OSA) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR-1112-AGPAP-MS
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): REMStar auto A-Flex
  Interventions: Device: REMstar Auto A-Flex
- Group 2 (Experimental): modified REMstar Auto A-Flex with AGPAP
  Interventions: Device: modified REMstar Auto A-Flex with AGPAP

INTERVENTIONS:
Device: REMstar Auto A-Flex — Standard CPAP
  Other Names: Philips Respironics System One
  Arms: Group 1
Device: modified REMstar Auto A-Flex with AGPAP — Modified device -Software upgrade to GP 12
  Other Names: Philips Respironics System One
  Arms: Group 2

SUMMARY:
Although positive airway pressure (PAP) is a highly effective treatment for sleep apnea, adherence to therapy remains an obstacle. Automated Graduated CPAP (AGPAP), also know as EZ-start, is an extended duration ramp, where the patient receives pressure below their prescription during an acclimation phase. The algorithm gradually increases pressure to therapy level based on usage. The aim of this study was to determine the effectiveness of the AGPAP acclimation period and its impact on short term adherence.

DETAILED DESCRIPTION:
Even though CPAP is highly effective in treating sleep apnea, adherence to CPAP therapy remains the largest single obstacle to the successful resolution of sleep-disordered breathing in OSA patients. It has been estimated that up to 50% of patients who have been prescribed CPAP for Obstructive Sleep Apnea (OSA) are not using the treatment one year later. A myriad of possible causes for low compliance rates have been proposed and examined in previous studies. These include race, gender, education level, income, bed-partner's sleep quality, mask discomfort, continuity of care, nasal irritation, discomfort due to elevated expiratory pressure, and level of daytime sleepiness.

Therefore, many investigators have proposed new methods and approaches to help deal with these problems. Interventions have ranged from people-centric approaches using intensive CPAP education and follow-up programs, to device modifications using features such as a ramp, C-FLEX®, BiLevel therapy, and heated humidification.

In this study. The aim of this study was to determine the effectiveness of the Automated Graduated CPAP (AGPAP), also know as EZ-start acclimation period, and its impact on short term adherence

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with OSA (last 12 weeks)
* Prescribed continuous positive airway pressure (CPAP) pressure ≥ 10 cmH2O
* Willing and able to provide informed consent
* Able to follow instructions

Exclusion Criteria:

* Participation in another interventional research study within the last 30 days
* Major controlled or an uncontrolled medical condition such as congestive heart failure, neuromuscular disease, renal failure, cancer, chronic obstructive pulmonary disease (COPD), respiratory failure or insufficiency, or patients requiring oxygen therapy (as determined by self-report and reviewed by the study PI.)
* Prior PAP prescription, use, or any prior OSA treatment, excluding split-night or titration PAP exposure.
* Prescribed BiLevel therapy
* Presence of untreated, non-OSA related sleep disorders (e.g. moderate to severe restless legs (PLMAI ≥ 20) or insomnia)
* History of an automobile accident or near accident in the last 12 months due to sleepiness.
* Severe oxygen desaturation on the PSG (Sa02 < 70% for 10% of the diagnostic PSG study).
* Surgery of the upper airway, nose, sinus, or middle ear within the past 90 days
* Regular use (>3 nights per week) of sleeping pills or stimulants.
* Currently working a night shift or rotating day/night shift.
* Unwillingness to try PAP at home.
* Presence of tracheostomy

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lankford, PhD, Principal Investigator — Sleep Disorders Center of Georgia
Locations (5):
- United States (5):
  - Delta Waves Sleep Disorder and Research Center, Colorado Springs, Colorado
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Clayton Sleep Institute, St Louis, Missouri
  - Clinilabs, Inc., New York, New York
  - Sleep Therapy and Research Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 123 | 118
Completed | 101 | 82
Not Completed | 22 | 36
Not completed — Withdrawal by Subject | 19 | 13
Not completed — protocol deviation | 3 | 23

BASELINE CHARACTERISTICS:
Population: 241 participants were enrolled in the trial and randomized, 123 in group 1 and 118 in group 2. there were 3 protocol deviations in group 1 and 23 deviations in group 2. data from these participants were excluded from the final analysis as per the statistical plan, and an intention to treat analysis was performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 120 | 115 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (10.5) | 46.2 (11.0) | 47.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 42 | 91
  Male | 71 | 73 | 144
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120 | 115 | 235
Apnea-hypopnea index (AHI) [Mean (Standard Deviation); unit: events/hour] | 44.6 (34.6) | 42.2 (31.1) | 43.4 (32.9)
CPAP Prescription [Mean (Standard Deviation); unit: cmH2O] | 12.1 (2.1) | 12.3 (2.2) | 12.2 (2.2)
Functional Outcomes Sleep Questionnaire (FOSQ) (quality of life questionnaire [Mean (Standard Deviation); unit: units on a scale] — Functional Outcomes Sleep Questionnaire (FOSQ) is a self-administered instrument designed to assess the impact of excessive sleepiness on daytime function and to quantify improvement after treatment. It contains 30 items divided into 5 subscales: Activity level, vigilance, intimacy and sexual relationships, general productivity, and social outcome. The patient rates the difficulty of performing a given activity on a 4-point scale (no difficulty to extreme difficulty)
  A mean score is calculated for each scale ranging from 0 (maximum functional impact) to 24 (no functional impact).
  units on a scale | 2.9 (0.6) | 2.8 (0.7) | 2.8 (0.6)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score can range from 0 to 24. The higher the ESS score, the higher is the overall 'daytime sleepiness'.
  units on a scale | 12.2 (4.6) | 11.6 (5.1) | 11.9 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: CPAP Adherence
Description: Device usage (hours per night)
Time Frame: 3 months
Population: 241 participants were enrolled in the trial and randomized, group 1 = 123 and group 2 = 118. There were 3 protocol deviations in group 1 and 23 deviations in group 2. Data from these participants were excluded from the final analysis as per the statistical plan, and an intention to treat analysis was performed.
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 120 | 95
hours per night | 3.6 (2.5) | 4.0 (2.3)

2. Secondary Outcome: Functional Outcome Sleep Quality (FOSQ)
Description: Functional Outcomes Sleep Questionnaire (FOSQ) is a self-administered instrument designed to assess the impact of excessive sleepiness on daytime function and to quantify improvement after treatment. It contains 30 items divided into 5 subscales: Activity level, vigilance, intimacy and sexual relationships, general productivity, and social outcome. The patient rates the difficulty of performing a given activity on a 4-point scale (no difficulty to extreme difficulty) A mean score is calculated for each scale ranging from 0 (maximum functional impact) to 24 (no functional impact).
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1- Standard CPAP: REMStar auto A-Flex
  REMstar Auto A-Flex: Standard CPAP
- Group 2 -AGPAP: modified REMstar Auto A-Flex with AGPAP
  modified REMstar Auto A-Flex with AGPAP: Modified device -Software upgrade to GP 12
Arm/Group | Group 1- Standard CPAP | Group 2 -AGPAP
Number analyzed (Participants) | 120 | 115
units on a scale | 3.35 (0.68) | 3.25 (0.64)

3. Secondary Outcome: Daytime Sleepiness as Measured by the Epworth Sleepiness Scale
Description: Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score can range from 0 to 24. The higher the ESS score, the higher is the overall 'daytime sleepiness'.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1- Standard CPAP | Group 2 -AGPAP
Number analyzed (Participants) | 120 | 115
units on a scale | 8.05 (4.45) | 8.27 (4.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the device trial period, e.g. 3 months
Arm/Group | Group 1- Standard CPAP | Group 2 -AGPAP
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/115
Serious Adverse Events (participants affected / at risk) | 2/120 | 1/115
Other Adverse Events (participants affected / at risk) | 30/120 | 33/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- Standard CPAP (N=120) | Group 2 -AGPAP (N=115)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization (Cardiac disorders) | 1 (1) | 0 (0) — Participant 404 was hospitalized with complaints of dizziness and light-headed. The report obtained from the Hospital lists subconjunctival hemorrhage, severe uncontrolled hypertension, and uncontrolled diabetes as the main findings
Bipolar manic episode (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1- Standard CPAP (N=120) | Group 2 -AGPAP (N=115)
Dry mouth (General disorders) | 5 (5) | 4 (4)
Aerophagia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Cold/flu symptoms (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 19 (24)
Bronchites/asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hand fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Broken & casted R carpal, 5th digit
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Ankle swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upset stomach and diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (4)
cracked dental implant (General disorders) | 0 (0) | 1 (1)
Dry, Stuffy Nose or Nosebleeds, skin irritation (Reproductive system and breast disorders) | 11 (11) | 4 (4) — These are common side effects of CPAP therapy. https://www.sleepassociation.org/sleep-apnea/cpap-treatment/cpap-side-effects/
Worsening of hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
MRSA in armpit (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No